CLINICAL TRIAL: NCT06372704
Title: Urinary Incontinence After Radical Prostatectomy Surgery is a Common Condition That Negatively Affects Daily Life. This Study Aimed to Evaluate the Efficacy and Safety of High-intensity Focused Electromagnetic Technology Used Therapeutically in Patients With Urinary Incontinence After Radical Prostatectomy. Our Study Has Shown That High-intensity Focused Electromagnetic Technology Can Safely and Effectively Treat Male Patients Suffering From Urinary Incontinence After Prostatectomy. In Addition, no Major Side Effects Were Observed in Patients After Treatment
Brief Title: Is the HIFEM Procedure an Effective Treatment for Men With Post-prostatectomy Incontinence?
Acronym: HIFEM for PPI
Status: Completed | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Ibrahim Untan, Deputy Chief Physician, Kirsehir Ahi Evran Universitesi
Other Study IDs: 2024/72
Record Dates: First submitted 2024-04-09; First posted 2024-04-18 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Prostate Cancer; Incontinence; Pelvic Floor Muscle Weakness
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- post prostatectomy incontinence: Twenty-seven patients who underwent radical prostatectomy with a mean age of 67.90 ± 3.40, and who had continuous UI complaints, were included in the study.
  Interventions: Device: HIFEM

INTERVENTIONS:
Device: HIFEM — All patients had a total of 6 sessions lasting 28 minutes, twice a week, sitting on an electromagnetic chair (BTL EMSELLA®, BTL Industries Inc, Boston, MA, USA).

SUMMARY:
Urinary incontinence after radical prostatectomy surgery is a common condition that negatively affects daily life. Patients often experience discomfort due to urine leakage and the resulting need to use pads daily. This study aimed to evaluate the efficacy and safety of high-intensity focused electromagnetic technology used therapeutically in patients with urinary incontinence after radical prostatectomy.

DETAILED DESCRIPTION:
Patients who underwent radical prostatectomy and who had continuous UI complaints, were included in the study. Informed consent forms were obtained from all volunteer patients before the procedure. Data was collected pre- and post-treatment. All patients had a total of 6 sessions lasting 28 minutes, twice a week, sitting on an electromagnetic chair (BTL EMSELLA®, BTL Industries Inc, Boston, MA, USA). According to the procedure, all patients remained fully clothed throughout the entire process. To ensure adequate PFM stimulation, the operator confirmed the patient's chair posture throughout the treatments and adjusted the intensity of stimulus as high as tolerated by the patient, usually at 100%. Ensuring the correct positioning is crucial for maximizing therapy effectiveness, so the therapist supervised the subject's posture and confirmed it using the device's positioning system to attain the best possible PFM contractions. Men with pacemakers, metal implants in the spinal cord, blood circulation disorders, fever, and tumors were excluded from the study.

The International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) was employed to evaluate each patients' continence. The questionnaire comprises three inquiries aimed at measuring how often leakage occurs, the volume of urine leaked, and the extent of disruption to daily activities. Scores on the questionnaire range from 0 (indicating no disruption) to 21 (representing significant involuntary urination affecting the individual's quality of life). A minimum of a 50% overall enhancement in the total score was anticipated(10). Participants were requested to mark the provided responses that applied to their situation, and alterations in their responses over time were assessed. Regarding the quality of life for the patient, the utilization of absorbent pads (per 24-hour cycle) was tracked using a questionnaire specifically designed for pad usage. Data on the primary outcome were collected before the first therapy, upon completion of the sixth therapy session, and at the first-month follow-up. Adverse events were monitored throughout the entire study. The assessment of observed side effects included the following in the treated area: muscle pain, temporary muscle spasms, temporary joint or tendon pain, local redness, or skin redness. The results were analyzed for statistical significance. H0 (null hypothesis) was formulated as follows: "The treatments did not make any difference in the patients' scores." To evaluate the significance of differences caused by treatments (alternative hypothesis), Student's paired t-test and Wilcoxon signed rank test were used if the sample size was small, the significance level was set at p = 0.05. A sample size of 27 individuals was considered sufficient to demonstrate clinically significant improvement for this single-arm retrospective study. The potential relationship between the measured variables was confirmed using the Pearson correlation coefficient (p = 0.05).

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent radical prostatectomy
* patients who had continuous UI complaints

Exclusion Criteria:

* Men with pacemakers, metal implants in the spinal cord, blood circulation disorders, fever, and tumors

Ages: 63 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Twenty-seven patients who underwent radical prostatectomy with a mean age of 67.90 ± 3.40, and who had continuous UI complaints, were included in the study.
Study Population: Patients who underwent radical prostatectomy with a mean age of 67.90 ± 3.40, and who had continuous UI complaints, without pacemakers, metal implants in the spinal cord, blood circulation disorders, fever, and tumors.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
This study demonstrated the safe and effective use of HIFEM technology to prevent PPI by strengthening the pelvic floor muscles in a variety of patients. | One month.
  The average International Consultation on Incontinence Questionnaire-Short Form score was calculated before and after the treatment. Their average "pads used per day" was calculated before and after the treatment. The scores and pads' numbers were compared statistically.

CONTACTS AND LOCATIONS:
Locations (1):
- İbrahim Üntan, Kirşehi̇r, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided